CLINICAL TRIAL: NCT05473312
Title: Women Supporting Women Using Local Solutions to Improve Infant and Young Child Feeding and Care Practices in Punjab, Pakistan
Brief Title: Women Supporting Women to Improve Infant and Child Feeding Practices
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: University of British Columbia (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr Sajid Bashir Soofi, Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IYCF Study
Record Dates: First submitted 2022-04-12; First posted 2022-07-25 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Undernutrition; Healthy Nutrition; Health Behavior; Health Knowledge, Attitudes, Practice; Child Malnutrition; Child Rearing; Health Care Seeking Behavior
MeSH Terms: conditions — Malnutrition; Health Behavior; Behavior; Child Nutrition Disorders; Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 1. Community Sensitization
  2. 28-day behaviour practice (Positive Deviance (PD) /Hearth sessions plus home practice)
  3. Supplemental Print Information
  Interventions: Behavioral: Community Sensitization; Behavioral: 28-day PD/Hearth Sessions; Behavioral: Supplemental Print Information
- Control (No Intervention): Control households will continue with usual practices.

INTERVENTIONS:
Behavioral: Community Sensitization — One event will be developed and delivered for households in each cluster area. Approach and content will be informed by the formative research and CAC input (may include drama and nutrition fairs).
  Arms: Intervention
Behavioral: 28-day PD/Hearth Sessions — Mothers will come together in a home-like setting to rehabilitate their malnourished child (8 dyads/Hearth), learn and practice new feeding and childcare behaviours (during Covid-19: 4 dyads/Hearth). Curriculum and activities will be informed by CAC, CORE Guide and formative research. Two female facilitators will demonstrate, encourage, convey key messages and guide practices.
  Arms: Intervention
Behavioral: Supplemental Print Information — The content will be informed by the formative research and CAC, will reinforce Hearth messages, and be adapted for each gender group. Material will be locally produced, engaging, user friendly, and target an illiterate audience (i.e. culturally relevant images with minimal text).
  Arms: Intervention

SUMMARY:
Undernutrition in the first 2 years of life is the largest preventable cause of death before age 5. Among those who survive, stunting before age two leaves millions with lifelong physical and cognitive deficits, which are difficult to compensate for later in life. Pakistan is home to the second largest number of stunted children in South Asia. The primary goal of this study is to rehabilitate moderately malnourished children aged 7-23 months and enable mothers to sustain this healthy growth at home by changing their infant and young child feeding (IYCF) practices, child care, hygiene and health-seeking behaviours.

DETAILED DESCRIPTION:
Background and Rationale:

Undernutrition in the first 2 years of life is the largest preventable cause of death before age 5. Among those who survive, stunting before age two leaves millions with lifelong physical and cognitive deficits, which are difficult to compensate for later in life. Pakistan is home to the second largest number of stunted children in South Asia. COVID-19 is projected to increase the prevalence of child malnutrition by almost 14% in the coming year, the majority of which will be in low-middle income countries (LMICs) like Pakistan. In the last two decades, there has been a little reduction in the prevalence of child undernutrition in Pakistan compared to other LMICs. With four in ten children under 5 years of age stunted, one in three underweight, and one in five wasted, Pakistan is a priority country for action to improve infant and young child feeding (IYCF) and caring practices. We will identify uncommon but successful (i.e. Positive Deviant -PD) IYCF behaviours practiced by local mothers of well-nourished children from economically disadvantaged homes, and transfer these practices to mothers with undernourished children who are equally disadvantaged in the wider community.

Goals: To rehabilitate moderately malnourished children aged 7-23 months and enable mothers to sustain this healthy growth at home by changing their IYCF practices, child care, hygiene and health-seeking behaviours.

Hypothesis: A higher proportion of children in the intervention compared to the control group will experience an average weight gain of 400g/month in the first 4 months of the intervention.

Objectives:

1. Understand local perceptions, experiences, cultural norms around IYCF practices and care,
2. Discover demonstrably successful IYCF behaviours and strategies using local resources,
3. Develop and implement a culturally appropriate and context specific intervention, and
4. Evaluate the intervention.

Approaches: This population health research will take place in two rural communities (tehsils) of Rahim Yar Khan District, Punjab, Pakistan. The tehsils will be randomly selected to either control or intervention. A community-based approach is being used to engage the community in planning, development, implementation and evaluation. Study activities will involve (1) formative research (focus groups and household inquiry/observation) to identify PD IYCF practices, (2) development of a behaviour change intervention informed by the formative research data, (3) delivery of the intervention to mothers and fathers of malnourished children using community sensitization events, print information, and home-like settings for mothers to learn and practice the new behaviours, and (4) a quasi-experimental design using focus groups, household surveys, and children's growth patterns to evaluate the intervention.

Expertise: Our research team includes Canadian and Pakistani experts in community-based research, global health, behaviour change, qualitative and quantitative methods, and child nutrition, with a deep understanding of the community's beliefs concerning health and nutrition.

Expected Outcomes: The project will strategically position our team to guide efforts in Pakistan to improve undernutrition, with the potential to expand this work to other LMICs where our team is affiliated, such as Afghanistan and Uganda. This proposal is aligned with CIHR's mandate to advance global health research that addresses health inequities in LMICs.

ELIGIBILITY:
Inclusion Criteria:

* Households with a moderately malnourished child (Index child) 7-9 month of age and both parents consenting using thumbprint or written signature (one dyad/household).

Exclusion Criteria:

* Any disability that precludes providing informed consent, transient, < 18 yrs (legal consent age).

Ages: 7 Months to 9 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 350 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Child weight | Day 1 of each Hearth/home cycle
  Child weight measurement in kilograms
Child weight | Day 14 of each Hearth/home cycle
  Child weight measurement in kilograms
Child weight | Day 28 of each Hearth/home cycle
  Child weight measurement in kilograms
Child weight | Monthly for a total of 12 months
  Child weight measurement in kilograms

SECONDARY OUTCOMES:
Child length | Day 1 of each Hearth/home cycle
  Child length measurement in centimeters
Child length | Day 14 of each Hearth/home cycle
  Child length measurement in centimeters
Child length | Day 28 of each Hearth/home cycle
  Child length measurement in centimeters
Child length | Monthly for a total of 12 months
  Child length measurement in centimeters
Prevalence of infant and young child feeding knowledge and practices | At baseline
  Infant and young child feeding knowledge and practices will be measured using household survey questionnaire
Change in infant and young child feeding knowledge and practices | At 6 months
  Infant and young child feeding knowledge and practices will be measured using household survey questionnaire
Change in infant and young child feeding knowledge and practices | At 12 months
  Infant and young child feeding knowledge and practices will be measured at using household survey questionnaire
Prevalence of child care knowledge and practices | At baseline
  Child care knowledge and practices will be measured using household survey questionnaire
Change in child care knowledge and practices | At 6 months
  Child care knowledge and practices will be measured using household survey questionnaire
Change in child care knowledge and practices | At 12 months
  Child care knowledge and practices will be measured using household survey questionnaire
Prevalence of hygiene knowledge and practices | At baseline
  Hygiene knowledge and practices will be measured using household survey questionnaire
Change in hygiene knowledge and practices | At 6 months
  Hygiene knowledge and practices will be measured using household survey questionnaire
Change in hygiene knowledge and practices | At 12 months
  Hygiene knowledge and practices will be measured using household survey questionnaire
Prevalence of health-seeking knowledge and practices | At baseline
  Health-seeking knowledge and practices will be measured using household survey questionnaire
Change in health-seeking knowledge and practices | At 6 months
  Health-seeking knowledge and practices will be measured using household survey questionnaire
Change in health-seeking knowledge and practices | At 12 months
  Health-seeking knowledge and practices will be measured using household survey questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University Reseach Office, Rahim Yar Khan, Pakistan

IPD SHARING:
Plan to Share IPD: No